CLINICAL TRIAL: NCT03674918
Title: How to Reliably Diagnose Arterial Hypertension: Lessons From 24h Blood Pressure Monitoring.
Brief Title: Reliable Hypertension Diagnosis Based on 24 ABPM
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Principal Investigator, Hasselt University
Other Study IDs: 24 ABPM001
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- persons with arterial hypertension: patients referred to consultation cardiology for hypertension. They get a 24 h blood pressure monitoring to define the exact mean arterial blood pressure
  Interventions: Diagnostic Test: 24 h ambulatory blood pressure measurements

INTERVENTIONS:
Diagnostic Test: 24 h ambulatory blood pressure measurements — 24 h ambulatory blood pressure measurements : an ambulatory 24 h blood pressure device that automatically measures blood pressure every 15 minutes is given to the patient for 24 h

SUMMARY:
24 h blood pressure monitoring can help to define which is the optimal timing and frequency of measurements

DETAILED DESCRIPTION:
Hypertension is a common condition in modern society. As blood pressure fluctuates with time, a single blood pressure measurement is useless to diagnose hypertension. Nevertheless, a questionable not well-defined number of measurements still is often used for this purpose. Diagnosis and therapeutic control of hypertension are therefore suboptimal. This study's objective is to determine the number and timing of measurements needed to give a trustworthy approximation of an individual's average blood pressure. Therefore, 24 h ambulatory blood pressure measurements were retrospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 70 per cent of valid measurements

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Arterial hypertension, HBPM, 24h ABPM, optimal diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Timing of measurement | day 1
  9:00-13:00 - 13:00-17:00 - 17:00 - 21:00: there intervals were analyzed to assess the predictive value of each interval compared with the overall daytime diagnosis of hypertension.

SECONDARY OUTCOMES:
The correct number of measurements | day 1
  Within the intervals, the correct number of measurements needed to diagnose hypertension will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Caro Brenard, student, Study Chair — University of Leuven; Vincent Raymaekers, student, Study Chair — Universiteit Antwerpen; Paul Dendale, prof. dr., Principal Investigator — Hasselt University; Ines Frederix, dr. MD, Study Director — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium